CLINICAL TRIAL: NCT01809574
Title: The Role of Rheumatological Evaluation in the Management of Patients With Interstitial Lung Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 225-12-MMC
Record Dates: First submitted 2013-03-10; First posted 2013-03-12 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2013-10

CONDITIONS: Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis; Connective Tissue Disease
Keywords: Interstitial lung disease; Idiopathic pulmonary fibrosis; Connective tissue disease
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis; Connective Tissue Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We hypothesized that the multi-disciplinary assessment of interstitial lung disease patients would lead to a more accurate diagnosis and consequently alterations in treatment regimens that may lead to improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old
* ILD according to ATS/ERS guidelines
* Signed inform consent

Exclusion Criteria:

* Previous lung surgery
* Other significant systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients that will refer to the pulmonary outpatient or inpatients department for evaluation due to ILD will be included
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The number of patients with collagen related pulmonary fibrosis that are diagnosed by Rheumatologists compared to Pulmonologists. | two years

CONTACTS AND LOCATIONS:
Overall Officials: David Shitrit, Dr, Principal Investigator — Head of Pulmonary departmant, Meir Medical Center.
Locations (1):
- Meir Medical Center, Kfar Saba, Israel, Israel